CLINICAL TRIAL: NCT04927026
Title: "Where-there-is-no-psychiatrist Integrated Personal Therapy" Among Community-Dwelling Older Adults: Feasibility Randomized Controlled Trial
Brief Title: "Where-there-is-no-psychiatrist Integrated Personal Therapy" Among Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Shefaly Shorey, Principal investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A17-2003-B
Record Dates: First submitted 2021-06-01; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Older Adults; Mental Health; Mindfulness; Solution-focused Brief Therapy
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Where-there-is-no-psychiatrist Integrated Personal Therapy (WIPT) (Experimental): Solution-focused brief therapy (SFBT) involving psychoeducation and structured life review therapy, as well as mindfulness-based training
  Interventions: Behavioral: Where-there-is-no-psychiatrist Integrated Personal Therapy (WIPT)
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Where-there-is-no-psychiatrist Integrated Personal Therapy (WIPT) — The WIPT include weekly face-to-face group sessions including mindfulness-based training and solution focused brief therapy (SFBT) involving psychoeducation and structured life review therapy catered to the personal needs of the participants.
  Arms: Where-there-is-no-psychiatrist Integrated Personal Therapy (WIPT)

SUMMARY:
The World Health Organization (WHO) reported that approximately 15% of adults aged 60 and above suffer from some form of mental disorder, with one of the most common neuropsychiatric disorders being depression. Similar trends are seen in Singapore where 11.4% of the older adults aged 65 and above had depressive symptoms. Another population survey conducted among elderly in Singapore showed that elderly with subsyndromal depression (SSD) were similar to or worse than elderly with Major Depressive Disorder (MDD). However being a multi-ethnic Asia society the mental conditions such as depression and anxiety are seen as taboo topics to be discussed more so to seek help or treatment for these conditions in Singapore. Additionally scarcity of trained psychiatrists and work load of these trained professionals in the acute care settings make it difficult to reach these needy older adults. Hence, it is imperative to support the needs of this group of community dwelling older adults to ensure that their emotional wellbeing, and their condition do not progress to MDD. As such, this is the first of its kind study that will evaluate the effectiveness of solution focused brief therapy delivered by the lay mindfulness practitioner and the nurses.

If the pilot intervention is found to be feasible and effective, the large scale community trial will be planned to reach to more elderly in Singapore to help them age in a dignified way. In addition, other countries that do not involve lay mindfulness practitioners and nurses to provide integrated personal therapy in the community may benefit from this study as well.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged between 60-95 years old
* Able to understand and speak either English and/or Mandarin
* Able to attend at least 80% (five out of seven sessions) of the intervention sessions
* Have subsyndromal depression (obtained a score between one and five on the Geriatric Depression Scale) and/or subsyndromal anxiety (obtained a score between three and 10 on the Geriatric Anxiety Scale)

Exclusion Criteria:

* Older adults aged between 60-95 years old without subsyndromal depression and/or subsyndromal anxiety
* Older adults aged between 60-95 years old who could not understand or speak either English and/or Mandarin.
* Older adults aged between 60-95 years old who were unable to attend at least 80% (five out of seven sessions) of the intervention sessions.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression | Prior to start of intervention
  Measured using Geriatric Depression Scale. 15-item scale where participants select either "Yes" or "No" in response to 15 statements. The maximum score that could be obtained was 15 points; a high score on the scale indicates severe depressive symptoms.
Symptoms of depression | 3 months post-recruitment
  Measured using Geriatric Depression Scale. 15-item scale where participants select either "Yes" or "No" in response to 15 statements. The maximum score that could be obtained was 15 points; a high score on the scale indicates severe depressive symptoms.
Symptoms of depression | 6 months post-recruitment
  Measured using Geriatric Depression Scale. 15-item scale where participants select either "Yes" or "No" in response to 15 statements. The maximum score that could be obtained was 15 points; a high score on the scale indicates severe depressive symptoms.
Symptoms of anxiety | Prior to start of intervention
  Measured using Geriatric Anxiety Inventory. 20-item scale where participants select either "Agree" or "Disagree" to assess the anxiety symptoms in older adults. The maximum score that could be obtained was 20 points; a high score indicates more anxiety symptoms.
Symptoms of anxiety | 3 months post-recruitment
  Measured using Geriatric Anxiety Inventory. 20-item scale where participants select either "Agree" or "Disagree" to assess the anxiety symptoms in older adults. The maximum score that could be obtained was 20 points; a high score indicates more anxiety symptoms.
Symptoms of anxiety | 6 months post-recruitment
  Measured using Geriatric Anxiety Inventory. 20-item scale where participants select either "Agree" or "Disagree" to assess the anxiety symptoms in older adults. The maximum score that could be obtained was 20 points; a high score indicates more anxiety symptoms.

SECONDARY OUTCOMES:
Life satisfaction | Prior to start of intervention
  Measured using Satisfaction with Life Scale. 5-item scale that included a 7-point Likert scale (1 = "Strongly Disagree"; 7 = "Strongly Agree"). The maximum score that could be obtained was 35 points; a high score indicates high level of satisfaction with life.
Life satisfaction | 3 months post-recruitment
  Measured using Satisfaction with Life Scale. 5-item scale that included a 7-point Likert scale (1 = "Strongly Disagree"; 7 = "Strongly Agree"). The maximum score that could be obtained was 35 points; a high score indicates high level of satisfaction with life.
Life satisfaction | 6 months post-recruitment
  Measured using Satisfaction with Life Scale. 5-item scale that included a 7-point Likert scale (1 = "Strongly Disagree"; 7 = "Strongly Agree"). The maximum score that could be obtained was 35 points; a high score indicates high level of satisfaction with life.
Social connectedness in terms of friendship | Prior to start of intervention
  Measured using Friendship Scale. 6-item where participants had to select an answer out of the five options (1 = "Not at All"; 5 = "Almost Always"). The maximum score that could be obtained was 30 points; a high score indicates high level of social connectedness.
Social connectedness in terms of friendship | 3 months post-recruitment
  Measured using Friendship Scale. 6-item where participants had to select an answer out of the five options (1 = "Not at All"; 5 = "Almost Always"). The maximum score that could be obtained was 30 points; a high score indicates high level of social connectedness.
Social connectedness in terms of friendship | 6 months post-recruitment
  Measured using Friendship Scale. 6-item where participants had to select an answer out of the five options (1 = "Not at All"; 5 = "Almost Always"). The maximum score that could be obtained was 30 points; a high score indicates high level of social connectedness.
Quality of life | Prior to start of intervention
  Measured using World Health Organization Quality of Life-Older Adults module. 13-item scale where participants had to select an answer based on a 5-point rating scale (1 = "Not at All"; 5 = "Very Satisfied"). The maximum score was 65 points, and a high score indicates high quality of life.
Quality of life | 3 months post-recruitment
  Measured using World Health Organization Quality of Life-Older Adults module. 13-item scale where participants had to select an answer based on a 5-point rating scale (1 = "Not at All"; 5 = "Very Satisfied"). The maximum score was 65 points, and a high score indicates high quality of life.
Quality of life | 6 months post-recruitment
  Measured using World Health Organization Quality of Life-Older Adults module. 13-item scale where participants had to select an answer based on a 5-point rating scale (1 = "Not at All"; 5 = "Very Satisfied"). The maximum score was 65 points, and a high score indicates high quality of life.

OTHER OUTCOMES:
Cortisol in ng/ml | Prior to start of intervention
  Stress- and anxiety- related inflammatory outcomes. Collected in lithium heparin tubes
Cortisol in ng/ml | 6 months post-recruitment
  Stress- and anxiety- related inflammatory outcomes. Collected in lithium heparin tubes
Annexin-A1 in ng/ml | Prior to start of intervention
  Stress- and anxiety- related inflammatory outcomes. Collected in lithium heparin tubes
Annexin-A1 in ng/ml | 6 months post-recruitment
  Stress- and anxiety- related inflammatory outcomes. Collected in lithium heparin tubes
Interleukin-1-beta in pg/ml | Prior to start of intervention
  Stress- and anxiety- related inflammatory outcomes. Collected in lithium heparin tubes
Interleukin-1-beta in pg/ml | 6 months post-recruitment
  Stress- and anxiety- related inflammatory outcomes. Collected in lithium heparin tubes

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No